CLINICAL TRIAL: NCT05088512
Title: Preventive and Personalized Medicine (2021-2023)
Brief Title: The Role of Genetic Factors in the Development of Bronchial Asthma in the Kazakh Population
Status: Completed | Type: Observational
Sponsor: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Principal Investigator, Ildar Fakhradiyev, Project manager, Asfendiyarov Kazakh National Medical University
Other Study IDs: 1207
Record Dates: First submitted 2021-09-25; First posted 2021-10-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Bronchial Asthma; Genome Wide Association Studies
Keywords: Bronchial Asthma; Genome Wide Association Studies
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group:: Patients with bronchial asthma
  Interventions: Genetic: SNP analysis of the DNA
- Control group: Patients without bronchial asthma
  Interventions: Genetic: SNP analysis of the DNA

INTERVENTIONS:
Genetic: SNP analysis of the DNA — SNP analysis of the DNA obtained from peripheral blood sample

SUMMARY:
To research for a genetic marker of bronchial asthma, a single nucleotide polymorphism (SNP) analysis of DNA obtained from the peripheral blood of patients with bronchial asthma and normal control will be performed.

DETAILED DESCRIPTION:
Unrelated Kazaks subjects who have bronchial asthma were recruited in the current study. Genotyping for various SNP associated due to the linkage disequilibrium patterns is to be performed. Genotypes would be statistically compared between patients with bronchial asthma and normal control subjects free of bronchial asthma

ELIGIBILITY:
Inclusion Criteria:

* Persons with bronchial asthma confirmed by a doctor;
* The age of the patients is from 5 to 60 years;
* Persons of Kazakh nationality, whose paternal and maternal grandparents are Kazakhs.
* Persons who are able and willing to provide written informed consent;
* Persons capable and willing to comply with the research protocol;

Exclusion Criteria:

* Persons who, in the opinion of the researcher, are mentally or legally incapacitated, which prevents obtaining informed consent;
* Pregnant or lactating women;
* Tuberculosis of any localization in the active phase and in history;
* Severe and decompensated diseases of the liver and kidneys, cardiovascular system;
* Severe and decompensated course of endocrine diseases;
* Autoimmune diseases;
* Systemic diseases;
* Oncological diseases;

Ages: 5 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with bronchial asthma confirmed by a doctor
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-10-23 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
number of SNPs associated with bronchial asthma | 1 year
  Using SNPsto identify candidate genes associate with bronchial asthma

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakhstan, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided